CLINICAL TRIAL: NCT03112733
Title: Value of TFF3, SFRP4, Romo1 and NFKB as Serum Biomarkers in Diagnosis and Predicting Prognosis of Ovarian Cancers
Brief Title: Serum Biomarkers in Diagnosis and Predicting Prognosis of Ovarian Cancers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ilker Kahramanoglu (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor-Investigator, Ilker Kahramanoglu, MD, Gynecologic Oncology Fellow, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: 83045809-604.01.02; TAB-2017-22506 (Other Grant/Funding Number: Istanbul University, Scientific Research Projects)
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Endometrial Neoplasms; Ovarian Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with ovarian carcinoma: Serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-κB of patients with a presumed diagnosis of ovarian carcinoma will be determined prior to surgery.
  Interventions: Diagnostic Test: TFF3, SFRP4, Romo1, NFKB
- Control group: Serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-κB of women without any adnexal mass nor malignancy will be determined to compare with other groups.
  Interventions: Diagnostic Test: TFF3, SFRP4, Romo1, NFKB
- Benign adnexal mass: Serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-κB of women with an adnexal mass will be determined to compare with other groups.

INTERVENTIONS:
Diagnostic Test: TFF3, SFRP4, Romo1, NFKB — Blood samples of all participants will be collected.
  Groups: Control group; Patients with ovarian carcinoma

SUMMARY:
This study evaluates the usefulness of serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-κB as potential diagnostic and prognostic biomarkers in ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of epithelial ovarian carcinoma.

Exclusion Criteria:

* Patients with recurrence.
* Patients who received neoadjuvant chemotherapy or radiotherapy
* Presence of any secondary malignancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian carcinoma who will be operated in Cerrahpasa Medical Faculty, Division of Gynecologic Oncology will participate into the study. Additionally, women without any malignancy will participate as control group.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-Κb in discrimination of benign and malignant gynecologic disease | 2 days
  To measure serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-κB between groups and to identify a possible significant diagnostic marker

SECONDARY OUTCOMES:
Efficacy of serum levels of trefoil factor 3 (TFF3), secreted frizzled related protein 4 (sFRP-4), reactive oxygen species modulator 1 (Romo1) and nuclear factor (NF)-Κb in predicting overall survival and disease-free survival | 1 year
  To determine any relationship between prognosis of ovarian cancer and serum levels of four different biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Kahramanoglu, Principal Investigator — Istanbul University Cerrahpasa Medical Faculty; Macit Arvas, Study Chair — Istanbul University Cerrahpasa Medical Faculty; Fuat Demirkiran, Study Director — Istanbul University Cerrahpasa Medical Faculty; Tugan Bese, Study Director — Istanbul University Cerrahpasa Medical Faculty; Hasan Turan, Principal Investigator — Istanbul University Cerrahpasa Medical Faculty; Hafize Uzun, Study Director — Istanbul University Cerrahpasa Medical Faculty; Salvatore Giovanni Vitale, Study Director — University of Messina
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data may be shared with researchers planning to perform a metaanalysis.

REFERENCES:
- [Result] Lee SH, Lee JS, Lee EJ, Min KH, Hur GY, Lee SH, Lee SY, Kim JH, Lee SY, Shin C, Shim JJ, Kang KH, In KH. Serum reactive oxygen species modulator 1 (Romo1) as a potential diagnostic biomarker for non-small cell lung cancer. Lung Cancer. 2014 Aug;85(2):175-81. doi: 10.1016/j.lungcan.2014.05.023. Epub 2014 Jun 5. PMID 24951318
- [Result] Xu C, Zeng XH, Wang L, Tao SQ, Wu QX, Zhu P, Deng GH, Wang YM. sFRP-4, a potential novel serum marker for chronic hepatitis B-related hepatocellular carcinoma. Hepatobiliary Pancreat Dis Int. 2015 Apr;14(2):164-70. doi: 10.1016/s1499-3872(15)60352-6. PMID 25865689
- [Result] Nunes JJ, Pandey SK, Yadav A, Goel S, Ateeq B. Targeting NF-kappa B Signaling by Artesunate Restores Sensitivity of Castrate-Resistant Prostate Cancer Cells to Antiandrogens. Neoplasia. 2017 Apr;19(4):333-345. doi: 10.1016/j.neo.2017.02.002. Epub 2017 Mar 19. PMID 28319807
- [Result] Edfeldt K, Daskalakis K, Backlin C, Norlen O, Tiensuu Janson E, Westin G, Hellman P, Stalberg P. DcR3, TFF3, and Midkine Are Novel Serum Biomarkers in Small Intestinal Neuroendocrine Tumors. Neuroendocrinology. 2017;105(2):170-181. doi: 10.1159/000452891. Epub 2016 Nov 9. PMID 27829249